CLINICAL TRIAL: NCT03624790
Title: Phase I, Open Label, Inpatient Challenge Study of rRSV A/Maryland/001/11, a Human Respiratory Syncytial Virus Challenge Strain, Administered to Healthy Adult Volunteers
Brief Title: Inpatient Challenge Study of rRSV A/Maryland/001/11, a Human Respiratory Syncytial Virus Challenge Strain, Administered to Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIR 320
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: rRSV A/Maryland/001/11 (Experimental): Participants will receive a single dose of rRSV A/Maryland/001/11 at study entry (Day 0).
  Interventions: Biological: rRSV A/Maryland/001/11
- Cohort 2: rRSV A/Maryland/001/11 (Experimental): Participants will receive a single dose of rRSV A/Maryland/001/11 at study entry (Day 0).
  Interventions: Biological: rRSV A/Maryland/001/11

INTERVENTIONS:
Biological: rRSV A/Maryland/001/11 — 10^5 PFU; delivered intranasally

SUMMARY:
The purpose of this study is to evaluate the safety, infectivity and replication, and immunogenicity of a recombinant respiratory syncytial virus (rRSV A/Maryland/001/11) challenge virus administered intranasally to healthy adults.

DETAILED DESCRIPTION:
This study will evaluate the safety, infectivity and replication, and immunogenicity of a recombinant respiratory syncytial virus (rRSV A/Maryland/001/11) challenge virus administered intranasally to healthy adults.

Participants will be admitted to the inpatient isolation unit and will receive a single dose of 10^5 plaque forming units (PFUs) of rRSV A/Maryland/001/11, delivered intranasally on Day 0. Participants will be enrolled outside of the RSV season between April 1 and October 31.

Participants will remain in the inpatient isolation unit for a minimum of 8 days after the challenge and will be discharged after two RSV reverse transcription polymerase chain reaction (RT-PCR) results lower than 3 Log10 genome equivalents per mL of nasal wash.

Upon discharge from the inpatient unit, participants will attend outpatient visits on Days 10 (if previously discharged), 28, and 56. These study visits may include physical examinations, blood collection, and nasal washes. At 6 months, there will be a follow-up phone contact to assess for any new chronic conditions or serious health events/hospitalizations.

Volunteers in Cohort 1 received a dose of 10^5 PFU, consistent with similar RSV challenge studies done previously. Cohort 2 will be conducted as an extension of Cohort 1 to extend the safety and infectivity evaluation, and will also receive a single dose of 10^5 PFU rRSV A/Maryland/001/11 challenge.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults between 18 years and 50 years of age, inclusive.
* General good health, without significant medical illness, physical examination findings, or significant laboratory abnormalities as determined by the investigator.
* Demonstrates comprehension of the protocol procedures and knowledge of RSV illness by passing a written comprehension examination (pass grade greater than or equal to 70%).
* Available for the duration of the trial.
* Willingness to participate in the study and stay confined to the inpatient unit for the required duration as evidenced by signing the informed consent document.
* Participants with childbearing potential must agree to have used effective birth control methods beginning at least one month prior to challenge, and continuing with 'per label/fully effective use' for the chosen method for the duration of the study, from amongst these:

  * pharmacologic/hormonal contraceptives, including oral, parenteral, subcutaneous, and transcutaneous delivery;
  * condoms or diaphragm with spermicide;
  * intrauterine device;
  * absolute abstinence from heterosexual intercourse as a matter of normal preferred lifestyle;
  * or must be surgically sterile, or must be 50 years of age AND have had no menses at all for at least one full year.
  * All participants of childbearing potential must provide samples for urine and serum pregnancy testing prior to enrollment, prior to challenge, as well as a statement of menstrual history, at each study contact throughout the study, and report if they may be pregnant immediately.
* Willingness to refrain from blood and plasma donation for 1 year after study enrollment.
* Willingness to refrain from receiving licensed or investigational vaccines or other investigational products from the day of enrollment until Study Day 56.
* Willingness to follow admission and isolation requirements for the indicated duration per protocol.

Exclusion Criteria:

* Subject who was previously challenged with RSV in any study, or previously participated in an RSV vaccine study.
* Any subject who is pregnant or lactating OR planning to become pregnant in the timeframe that begins 30 days prior to the inoculation and ends 30 days after inoculation. Pregnancy is determined by a positive test for human chorionic gonadotropin (β-HCG test).
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies.
* Behavioral or cognitive impairment or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol.
* A history of asthma within the past 5 years, or a current diagnosis of asthma or reactive airway disease associated with exercise, seasonal hay fever or allergic rhinitis.
* Presence of any febrile illness or symptoms suggestive of a respiratory infection within 2 weeks prior to inoculation.
* Use of systemic or nasal steroid preparations or immunosuppressive drugs within 30 days prior to challenge. Topical steroid preparations are permitted.
* Inhaled bronchodilator or inhaled steroid use within the last year or use after upper respiratory tract infections within the last 5 years.
* Current or past (in the last 4 weeks) use of i.n. medications (including steroids, decongestants, or hormonal medications), or planning to use them within 28 days of study challenge
* Positive urine drug toxicology test for the presence of amphetamine, barbiturates, opiates, phencyclidine, benzodiazepines, methadone or cocaine metabolites.
* Evidence of current alcohol or illicit drug abuse or addiction.
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.
* History of anaphylaxis.
* Positive enzyme-linked immunosorbent assay (ELISA) and confirmatory tests for human immunodeficiency virus (HIV).
* Positive ELISA and confirmatory test (e.g., recombinant immunoblot assay) for hepatitis C virus (HCV).
* Positive hepatitis B virus surface antigen (HBsAg) by ELISA.
* Known immunodeficiency syndrome.
* Receipt of a live vaccine within 4 weeks or a killed vaccine within 2 weeks prior to inoculation with RSV challenge and planned receipt within 56 days after challenge.
* History of surgical splenectomy.
* Receipt of blood or blood-derived products (including immunoglobulin [Ig]) within 6 months prior to study inoculation.
* Current routine (at least once weekly) smoking or vaping of a tobacco product or marijuana.

  * The decision to exclude a potential subject is determined by medical history and a clinician's clinical judgment based on the physical examination.
* Receipt of any investigational vaccine or drug within 28 days prior or planned use within 56 days after study inoculation.
* Body mass index (BMI) less than 18.5 or greater than 37.5.
* Shared household, works closely with, or has routine contact with a child (children) less than 2 years of age or with immunocompromised individual(s), adults with significant cardiopulmonary disease, persons with significant asthma, institutionalized elderly or elderly with functional disability or any other individual that, in the judgment of the Principal Investigator (PI), might be at increased risk for complications if exposed to RSV.
* Any significant abnormality of the nose or nasopharynx, including recurrent epistaxis and including nasal or sinus surgery.
* History of Bell's palsy.
* Unwillingness to have nasopharyngeal (NP) swabs, nasal wash, or blood samples saved for future respiratory virus research.
* Serum RSV neutralizing antibody titers greater than or equal to 320.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Frequency of challenge virus-related solicited signs and symptoms | Measured through Day 56
  Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Severity of challenge virus-related solicited signs and symptoms | Measured through Day 56
  Graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Frequency of adverse events (AEs) | Measured through Day 56
  Graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Severity of AEs | Measured through Day 56
  Graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 2.1, March 2017
Number of participants infected with rRSV A/Maryland/001/11 challenge virus | Measured through Day 56
  Defined as recovery of challenge virus from nasal wash, and/or detection of virus in nasal wash by real-time reverse transcription polymerase chain reaction (rRT-PCR), and/or a greater than or equal to 2.5-fold rise in serum neutralizing antibody titer to RSV
Nasal wash virus titers of challenge virus shed | Measured through Day 56
  Measured by plaque titration and rRT-PCR
Number of days challenge virus was shed | Measured through Day 56
  Measured by plaque titration and rRT-PCR
Titer of serum immunoglobulin G (IgG) antibodies to the RSV F protein | Measured through Day 56
  Measured by enzyme-linked immunosorbent assay (ELISA)
Change in serum neutralizing antibody titer to RSV | Measured through Day 56
  Measured by plaque reduction assay

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Talaat, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03624790/ICF_000.pdf